CLINICAL TRIAL: NCT03425812
Title: Effects of Nonsteroidal Anti-Inflammatory Drugs (NSAIDs) in Recurrence of Spondyloarthritis (SPA) Patients After Remission：A Multicenter, Randomized, Controlled Study
Brief Title: Effects of Nonsteroidal Anti-Inflammatory Drugs in Recurrence of Spondyloarthritis Patients After Remission
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Collaborators: First Affiliated Hospital of Fujian Medical University (Other); Peking University Shenzhen Hospital (Other); Zhangzhou Affiliated Hospital of Fujian Medical University (Other); Quanzhou Orthopedic-traumatological Hospital of Fujian Traditional Chinese Medicine University (Unknown); Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20180101
Record Dates: First submitted 2018-01-19; First posted 2018-02-08 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Axial Spondyloarthritis
Keywords: Axial Spondyloarthritis; Anti-Inflammatory Drugs; Flare
MeSH Terms: conditions — Axial Spondyloarthritis | interventions — Anti-Inflammatory Agents, Non-Steroidal; Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Non- NSAIDS group (Experimental): To withdraw NSAIDS therapy
  Interventions: Drug: To withdraw NSAIDs therapy
- NSAIDS group (Active Comparator): To continue NSAIDS therapy
  Interventions: Drug: To continue NSAIDs therapy

INTERVENTIONS:
Drug: To withdraw NSAIDs therapy — NSAIDs therapy will be withdrew after washout period.
  Other Names: Non-NSAIDs; Break-off (on-demand) NSAID therapy; Break-off NSAID use (on-demand) group
  Arms: Non- NSAIDS group
Drug: To continue NSAIDs therapy — NSAIDs therapy will be continued.
  Other Names: NSAIDs; Regular (continuous) NSAID therapy; Regular (continuous) group
  Arms: NSAIDS group

SUMMARY:
The multicenter, randomized controlled trial is to investigate and evaluate the effect of NSAIDs therapy on recurrence in patients with axial spondyloarthritis;

DETAILED DESCRIPTION:
To investigate the recurrence rate in remission patients who withdraw NSAIDs therapy in axial spondyloarthritis;

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving informed consent and complying with the examination program of the protocol;
* Participants with axial SpA fulfilling the Assessment of Spondyloarthritis international Society 2009 (ASAS) axial SpA classification criteria;
* Participants must fulfill the criteria of maintaining remission of aSpA, defined as ASDAS<1.3；
* Participants must fulfill the criteria of remission of aSpA defined as ASDAS<1.3，then continuous to evaluate every four weeks for three times and ASDAS<1.3 each time.
* Laboratory results must fulfill following requirements: Hb≥85g/L；3.5×109/L≤WBC Count ≤10×109/L；Platelet count ≥ Normal lower limit; Liver function (ALT、TBIL) ≤Twofold of normal upper limit; Renal function (SCr) ≤Normal upper limit;
* The pregnancy test must be negative for women of childbearing age; Efficient contraception must be taken for both male and female participants during the trial period and within three months after the end of the trial.

Exclusion Criteria:

* Participants who previously have experienced allergic reactions to NSAIDs or sulfa-drugs;
* Participants who are intolerant of NSAIDs;
* Participants who are in active axSpA episodes;
* Participants with previous or currant ulcers and/or gastrointestinal conditions or bleeding in three months
* Participants who were in acute infection or acute attack of chronic infection during screening period;
* At the time of screening, participants who were in the acute stage of acute infection or chronic infection, and if the acute infection had improved, they could be re-screened.
* Participants who suffer from invasive fungal infections (e.g. histoplasma, coccidiosis's, candida, aspergillus, blastomyces, pneumocystis, etc.) within the first 6 months of screening; Or opportunistic bacterial infections (e.g. bacterial, viral or other infections, including Legionella and Listeria);
* Participants with other autoimmune diseases which are expected to influence the evaluation of experimental medications, such as inflammatory enteritis, psoriasis, uveitis, etc.
* Participants with previous or currant congestive heart failure, coronary heart disease, serious arrhythmia;
* Participants with severe, progressive, uncontrolled vital organ and systematic disorders, and other conditions that are considered inappropriate to participate in this trial;
* Participants with circumstances that may affect the compliance (e.g. prolonged travel or leave, planned relocation, mental illness, lack of motivation to participate, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2018-02-15 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2028-12-20 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with Ankylosing Spondylitis Disease Activity Score (ASDAS) active disease | From Week 0 (baseline) to Week24
  ASDAS active disease is defined as ΔASDAS-CRP≥0.9. The ASDAS is a composite disease activity outcome measure which combines patient reported back pain, duration of morning stiffness, patient global assessment of disease activity, patient assessment of peripheral joint pain and swelling and an acute phase reactant (CRP or ESR) as an objective measure of inflammation.

SECONDARY OUTCOMES:
Change in Patient global assessment of disease activity | From Week 0 (baseline) to Week24
  Participant rated instrument to measure participants' global assessment of disease activity on a 10 cm visual analogue scale, ranging from no activity to highest possible activity.
Change in total Back Pain | From Week 0 (baseline) to Week24
  Participants assessed the total back pain they had in the previous 1 week on a scale from 0 (no pain) to 10 (most severe pain).
Change in Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | From Week 0 (baseline) to Week24
  A numeric rating scale was used, for questions 1-5 (Fatigue, Spinal Pain, Joint pain or Swelling, Discomfort and Morning stiffness severity respectively) on a scale from 0 (none) to 10 (very severe). Question 6 (morning stiffness duration) was recorded on a scale of 0 (0 or more hours) to 10 (2 hours). To give the five major Ankylosing Spondylitis (AS) symptoms equal weighting, the average of the two scores relating to morning stiffness was taken. This averaged morning stiffness score was then summed with the remaining 4 questions, resulting in a composite score on a scale of 0-50, which was then divided by 5 to give the final BASDAI score on a scale of 0-10.
Change in Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) | From Week 0 (baseline) to Week24
  The BASFI is a participant's self-assessment represented as a mean (VAS; 0 to 10) of 10 questions, 8 of which relate to the participant's functional anatomy and 2 of which relate to a participant's ability to cope with everyday life. An increase along the scale indicates a worsening condition.
Change in Baseline in Bath Ankylosing Spondylitis Metrology Index (BASMI) | From Week 0 (baseline) to Week24
  BASMI is an objective measure of spinal mobility. The BASMI score is composed of 5 measures: cervical rotation, intermalleolar distance, modified Schober's test, lateral flexion and tragus to wall distance. Each measure was scored 0-2 (0=normal mobility, 2=severe reduction) to give a final score ranging 0 to 10.
Change in Short Form-36 Physical Component Summary (SF-36 PCS) | From Week 0 (baseline) to Week24
  The change from Baseline in Short Form-36 Physical Component Summary (SF-36 PCS)
Change in European Quality of Life-5 Dimensions (EQ-5D) Questionnaire | From Week 0 (baseline) to Week24
  The EQ-5D is an international, standardized, generic instrument for describing and valuing health status.In description part, health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. In evaluation part, the respondents evaluate their overall health status using the visual analogue scale (EQ-VAS).Visual analogue scale is the second part of the questionnaire, asking to mark health status on the day of the interview on a 20 cm vertical scale with end points of 0 and 100. There are notes at the both ends of the scale that the bottom rate (0) corresponds to " the worst health you can imagine", and the highest rate (100) corresponds to "the best health you can imagine".
Change in Chest Expansion | From Week 0 (baseline) to Week24
  Chest expansion, measured in cm, is defined as the difference in thoracic circumference during full expiration versus full inspiration, measured at the fourth intercostal space (nipple line). Chest expansion was measured for both maximum and minimum inhalation and the data presented below combined both the values.
Change in Maastricht Ankylosing Spondylitis Enthesitis Index (MASES) | From Week 0 (baseline) to Week24
  The MASES evaluation will be conducted at the designated study visits to assess the presence or absence of enthesitis at 13 different sites, noting the subjects' responses.
Change in Number of swelling and tendons affected by enthesitis | From Week 0 (baseline) to Week24
  An assessment of 44 swelling joints and 46 tendons joints will be done by physical examination at the designated study visits. Joint swelling will be classified as present (1), absent (0), replaced (9), or no assessment (NA).
Change in Blood samples: C-reactive protein (CRP) and Erythrocyte sedimentation rate(ESR) | From Week 0 (baseline) to Week24
  General and specific markers of inflammation. ESR will be evaluated at the site and expressed in mm/hg (1st hour).
Observation of relapse time after withdrawal of NSAIDs in remission patients | From Week 0 (baseline) to Week24
  ASDAS active disease is defined as ΔASDAS-CRP≥0.9
The difference of flare rate between different treatment groups | Week12 and Week24
  ASDAS active disease is defined as ΔASDAS-CRP≥0.9
The difference of flare rate between in patients with different sacroiliac joint grades on X-ray among different groups. | Week12 and Week24
  To grade radiographic sacroiliitis according to the New York criteria: grade0 normal; grade1 suspicious; grade2 minimal sacroiliitis; grade3 moderate sacroiliitis; grade4 ankylosis.
The difference of osteophyte formation between different groups on Modified Stoke ankylosing spondylitis spine score (mSASSS). | Week0 and Week24
  mSASSS focuses on the anterior vertebral body angles from the lower T12 endplate to the upper S1 endplate on a lateral radiograph. Each angle is scored 0 (normal), 1 (shiny corner sign, squaring, or sclerosis), 2 (enthesophyte), or 3 (bridging), so that the total score can range from 0 to 72.
Comparison of BASFI and BASMI scores between different groups | Week12 and Week24
  The BASFI is a participant's self-assessment represented as a mean (VAS; 0 to 10) of 10 questions, 8 of which relate to the participant's functional anatomy and 2 of which relate to a participant's ability to cope with everyday life. An increase along the scale indicates a worsening condition. BASMI is an objective measure of spinal mobility. The BASMI score is composed of 5 measures: cervical rotation, intermalleolar distance, modified Schober's test, lateral flexion and tragus to wall distance. Each measure was scored 0-2 (0=normal mobility, 2=severe reduction) to give a final score ranging 0 to 10.
Differences in MRI scores among different groups by SPARCC SSS method. | weeks-16, week 0, week 12 and week 24
  The SPARCC SSS method was developed based on semicoronal T1WSE sequences of the sacroiliac joints (SIJ). The transitional slice is identified by scrolling from anterior to posterior through the SIJ and viewing DICOM images depicting semicoronal slices through the joint. Scoring ranges are fat metaplasia (0-40), erosion (0-40), backfill (0-20), and ankylosis (0-20).
The difference of flare rate in patients with different MRI scores of sacroiliac joint. | Week0 and Week24
  MRI scores are measured by SPARCC SSS method.

CONTACTS AND LOCATIONS:
Overall Officials: Shi Guixiu, PhD, Study Director — The First Affiliated Hospital of Xiamen University
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zheng Q, Liu W, Huang Y, Gao Z, Wu Y, Wang X, Cai M, He Y, Chen S, Wang B, Liu L, Chen S, Huang H, Zheng L, Kang R, Zeng X, Chen J, Chen H, Chen J, Li Z, Shi G. Predictive Value of Active Sacroiliitis in MRI for Flare Among Chinese Patients with Axial Spondyloarthritis in Remission. Rheumatol Ther. 2021 Mar;8(1):411-424. doi: 10.1007/s40744-021-00279-y. Epub 2021 Feb 18. PMID 33598865